CLINICAL TRIAL: NCT02964000
Title: Adjunct Use of the Phoenix Thera-Lase for Treating Chronic Pain in Patients Taking Opioid-containing Medication on a PRN Basis
Brief Title: Phoenix Thera-Lase for Treating Chronic Pain in Patients Taking Opioid on a PRN Basis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phoenix Thera-lase Systems, LLC (Industry)
Responsible Party: Principal Investigator, Paul F. White, Professor, Phoenix Thera-lase Systems, LLC
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20162211
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Pain
Keywords: Pain; Low level laser therapy; Sham; Chronic Pain; Opioid; Physical activity; Quality of sleep
MeSH Terms: conditions — Pain; Chronic Pain; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low level 1 Watt (Active Comparator): The Phoenix Thera-Lase System will be on 1 watt while retaining appropriate "blinding" of both the operator and the patient.
  Treatments will be applied to the primary area of the body associated with pain for which analgesic (pain) medication is currently required.
  Each treatment session will last for 20-40 minutes.
  Interventions: Device: Low level 1 Watt
- Phoenix Thera-Lase System 42 (Experimental): The Phoenix Thera-Lase System will be on 42 watts while retaining appropriate "blinding" of both the operator and the patient.
  Treatments will be applied to the primary area of the body associated with pain for which analgesic (pain) medication is currently required.
  Each treatment session will last for 20-40 minutes.
  Interventions: Device: Phoenix Thera-Lase System 42
- Phoenix Thera-Lase System 74 (Experimental): The Phoenix Thera-Lase System will be on 74 watts while retaining appropriate "blinding" of both the operator and the patient.
  Treatments will be applied to the primary area of the body associated with pain for which analgesic (pain) medication is currently required.
  Each treatment session will last for 20-40 minutes.
  Interventions: Device: Phoenix Thera-Lase System 74

INTERVENTIONS:
Device: Low level 1 Watt — The Phoenix Thera-Lase System will be on 1 watt
  Other Names: 1 watt
  Arms: Low level 1 Watt
Device: Phoenix Thera-Lase System 42 — The Phoenix Thera-Lase System will be on 42 watts
  Other Names: 42 Watts
  Arms: Phoenix Thera-Lase System 42
Device: Phoenix Thera-Lase System 74 — The Phoenix Thera-Lase System will be on 74 watts
  Other Names: 74 Watts
  Arms: Phoenix Thera-Lase System 74

SUMMARY:
Hypothesis: Use of high level vs low level cold laser treatments will reduce chronic pain and the need for PRN opioid-containing analgesic medications.

Secondary Hypothesis: High level (vs low level) laser treatments will increase the patients level of physical activity and quality of sleep.

DETAILED DESCRIPTION:
Previous studies with low level laser therapy have reported beneficial effects on the level of pain in patients with a variety of chronic pain conditions.

We designed this controlled, double blind, randomized study to determine in the active laser group would have a reduction in the need for 'PRN pain medication'.

Screening Testing

1. Urine-toxicology screen.
2. Assessment of level of activity and range of motion and functional capacity evaluation for upper and/ or lower extremity.
3. Current drug history and use of analgesic medications including both opioid and or non-opioid analgesic medications.
4. Drug history and current medications along with non-traditional alternative treatments such as (e.g. acupuncture, massage, herbal treatments, etc.)

Protocol Outline After obtaining written informed consent, patients will be asked to complete all the pre-screening and "entry" questionnaires (e.g., SF-36).

11- point Verbal Rating Scale (VRS) for pain at rest and with physical activity (0= none to 10= severe), level of physical activity (0=inactive to 10= fully active), and quality of sleep (0=poor to 10=excellent).

Current analgesic [pain] medications both daily and PRN medications. Randomized into active (Phoenix Thera-Lase [ PTL]) or "Low level" PTL group using a computer generated random numbers table.

Treatment Sessions After obtaining written informed consent for participating in the study and signing the standard HIPPA forms, the patient will be asked to describe the location of their current pain symptoms.

Pre-treatment baseline assessments VRS for pain at rest and with physical activity (e.g. walking, climbing stairs) Kinesiology functional capacity evaluation (FCE) for upper and/ or lower extremities or low back (depending on location of pain).

Current opioid and non-opioid analgesic medication usage Clinical opioid withdrawal scale (COWS) at baseline (the COWS will be repeated at the end of the 1st, 2nd, and 3rd week of treatments).

Treatment sessions - Active or low level therapy for 20 - 40 min on Monday, Wednesday, and Friday for 3 weeks.

Post- treatment sessions VRS for pain at rest and with ambulation immediately after each treatment

After the end of 3-week treatment period Repeat pre-screening questionnaires. Kinesiology functional capacity evaluation (FCE) for upper and/ or lower extremities or low back (depending on location of pain).

Long-term Follow Up 30-days after the last treatment session, a standardized follow-up questionnaire will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* 25-65 years of age
* taking oral opiate-containing analgesic medication on a PRN
* patient with chronic pain related to an accident, injury or major surgery occurring within the past three years
* Patients with a potentially treatable pain condition
* Patient wiling to complete a daily diary for recording their pain score, activity level, quality of sleep and all pain-related medications for the three-week study period

Exclusion Criteria:

* Use of any opioid-containing pain medications for more than three years
* History of alcohol or drug abuse, or drug-seeking behavior
* Previous treatment for drug abuse in detox center or hospital
* Current psychiatric condition which require centrally- active medications
* Current excessive use of alcohol
* Any unstable medical conditions (e.g. coronary artery disease, hepato-renal or pulmonary disease)
* Patients not capable of consenting for themselves
* Pregnant women
* Women of child bearing potential not using acceptable birth control methods.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Reduce chronic pain | 1 month
reduce of opioid analgesic dosage. | one month

SECONDARY OUTCOMES:
Level of physical activity | 1 month
  It will be assessed with a questionnaire
Quality of sleep | one month
  It will be assessed with a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paul F White, PhD, MD, Principal Investigator — Phoenix Thera-Lase Systems
Locations (1):
- Phoenix Thera-Lase Systems, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes